CLINICAL TRIAL: NCT03386357
Title: Randomized Phase II Study of Immune Stimulation with Pembrolizumab and Radiotherapy in Second Line Therapy of Metastatic Head and Neck Squamous Cell Carcinoma (IMPORTANCE, Keynote-717, EudraCT NUMBER: 2017-002122-20 )
Brief Title: Radiotherapy with Pembrolizumab in Metastatic HNSCC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IMPORTANCE, Keynote-717
Record Dates: First submitted 2017-11-30; First posted 2017-12-29 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-10

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Open-label, Controlled, randomized trial
Masking Description: Open Label
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (pembrolizumab+RT) (Experimental): Pembrolizumab (200mg absolute, q3w) combined with radiotherapy (12x3Gy) of one, two or three metastases.
  Interventions: Combination Product: A (pembrolizumab+RT)
- B (pembrolizumab) (Active Comparator): Pembrolizumab (200mg absolute, q3w) without radiotherapy
  Interventions: Drug: B (pembrolizumab)

INTERVENTIONS:
Combination Product: A (pembrolizumab+RT) — Pembrolizumab (200mg absolute, q3w) combined with radiotherapy (12x3Gy) of one, two or three metastases. Only metastases that perspectively require radiotherapy will be treated. The irradiated tumor volume must be at least 10cm³. Radiotherapy of brain metastases is not allowed.
  Other Names: Keytruda + RT
  Arms: A (pembrolizumab+RT)
Drug: B (pembrolizumab) — Pembrolizumab (200mg absolute, q3w)
  Other Names: Keytruda
  Arms: B (pembrolizumab)

SUMMARY:
Randomized phase II study of immune stimulation with Pembrolizumab and radiotherapy in second line therapy of metastatic head and neck squamous cell carcinoma.

DETAILED DESCRIPTION:
This is an open-label, randomized, prospective, multicenter phase II clinical trial of pembrolizumab with or without local radiotherapy in patients with recurrent and/or metastatic HNSCC after progression to platinum-based therapy.

All patients will receive pembrolizumab 200mg absolute dose administered every third week. Patients in treatment arm A will receive radiotherapy of one, two or three metastases with a total tumor volume of at least 10cm³ intended to induce tumor cell death acting as an in situ vaccination. Radiotherapy will be performed conventionally fractioned with single doses of 3Gy to a total dose of 36Gy. There will be a strict time schedule. Radiotherapy will always start on Wednesday. After application of the third radiation dose (Friday) the patients will receive pembrolizumab. After an interruption of radiotherapy for two days (Saturday, Sunday), radiotherapy will be continued. Pembrolizumab will be continued on an every three week schedule until confirmed disease progression according to iRECIST criteria, unacceptable toxicity, patient's wish to stop therapy or a maximal treatment time of 12 months.

Tumor assessment will be performed every 9 weeks and will be evaluated according to iRECIST and RECIST. For each patient the same assessment method will be used throughout the study. Toxicity will be assessed according to CTCAE 4.0.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >18 years of age on day of signing informed consent.
3. Metastatic HNSCC (at least two distinct lesions: Lesion planned for radiotherapy with ≥10 ml tumor volume, or ≥3 lesions: 1 lesion planned for radiotherapy with ≥10 ml tumor volume or 2 lesions planned for radiotherapy with a cumulative tumor volume ≥10ml) OR Locally recurrent HNSCC not suitable for curative local treatment within or outside the previously irradiated tissue (at least two distinct lesions: Lesion planned for radiotherapy with ≥10 ml tumor volume, or ≥3 lesions: 1 lesion planned for radiotherapy with ≥10 ml tumor volume or 2 lesions planned for radiotherapy with a cumulative tumor volume ≥10ml).
4. Progression to first line platinum-based or any second/third line chemotherapy OR Progression within 6 months after platinum-based radiochemotherapy of locally advanced disease
5. Histological confirmation of HNSCC
6. Have at least one measurable lesion according to iRECIST that receives less than 10% of the prescribed dose of the irradiated lesion(s) (not considering doses from previous radiotherapy)
7. Have a performance status of 0-1 on the ECOG Performance Scale.
8. Demonstrate adequate organ function
9. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
10. Female subjects of childbearing potential (Section 5.7.2) must be willing to use an adequate method of contraception as outlined in Section 5.7.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
11. Male subjects of childbearing potential (Section 5.7.1) must agree to use an adequate method of contraception as outlined in Section 5.7.1- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

-

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., ≤ grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. History of (non-infectious) pneumonitis that required steroids, evidence of interstitial lung disease or active, non-infectious pneumonitis
11. Has an active infection requiring systemic therapy.
12. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
13. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
14. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
15. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent.
16. Has a known history of human immunodeficiency virus (HIV) (HIV 1/2 antibodies).
17. Has known active hepatitis B (e.g., HBsAg reactive) or hepatitis C (e.g., HCV RNA [qualitative] is detected).
18. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
19. Have a performance status of ≥2 on the ECOG Performance Scale.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2018-07-20 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Best response according to iRECIST criteria | Endpoint is the best response during pembrolizumab treatment (restaging every 9 weeks up to 12 months)
  Local radiotherapy will significantly improve the overall response rate according to iRECIST

SECONDARY OUTCOMES:
Response rate according to RECIST | restaging every 9 weeks up to 12 months
  RECIST 1.1 criteria
Assessment of target lesion | restaging every 9 weeks up to 12 months
  changes of the size of a (not irradiated) target lesion will be measured (%)
Assessment of the duration of response | restaging every 9 weeks up to 12 months
  The duration of the response will be evaluated in responding patients.
Assessment of the progression free survival | restaging every 9 weeks up to 12 months
  progression free survival (in months)
Assessment of the overall survival | restaging every 9 weeks up to 12 months
  Overall survival (in months)
Assessment of toxicity of the combination of pembrolizumab and radiotherapy | at every pembrolizumab administration (q3w) (up tp 12 months)
  Toxicity will be evaluated according to CTCAE 4.0

OTHER OUTCOMES:
Assessment of changes of the immunophenotype in peripheral blood after pembrolizumab without and with radiotherapy (longitudinal analysis) | week 1, at pembrolizumab administration 2, 4, 8, 12 and through study completion an average of 1 year
  Assessment of predictive value of PD-L1 in combination with tumor-infiltrating lymphocytes

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Fietkau, Prof., Study Chair — Universitätsklinikum Erlangen, Strahlenklinik; Wilfried Budach, Prof., Study Chair — University Düsseldorf; Markus Hecht, M.D., Principal Investigator — Universitätsklinikum Erlangen; Hausmann Jan, M.D., Study Chair — University Düsseldorf; Udo Gaipl, Prof., Study Chair — Universitätsklinikum Erlangen
Locations (7):
- Germany (7):
  - Bochum, St. Josef-Hospital, Abteilung für Hämatologie und Onkologie, Bochum
  - Dresden, Onkologische Gemeinschaftspraxis, Dresden
  - Düsseldorf, Universitätsklinikum, Klinik für Strahlentherrapie und Radiologische Onkologie, Düsseldorf
  - Erlangen, Universitätsklinikum Strahlenklinik, Erlangen
  - Frankfurt, Universitätsklinikum, Klinik für Strahlentherapie und Onkologie, Frankfurt
  - Homburg, Universitätsklinikum, Klinik für Strahlentherapie und Radioonkologie, Homburg
  - Regensburg, Universitätsklinikum, Klinik für Strahlentherapie, Regensburg

IPD SHARING:
Plan to Share IPD: No